CLINICAL TRIAL: NCT07086092
Title: Relationship Between Serum Markers and Motor Recovery and Ambulation in Post-stroke Patients: a Retrospective Analysis
Brief Title: Relationship Between Serum Markers and Motor Recovery and Ambulation in Post-stroke Patients
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, assistant professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-SK-11
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Biomarkers; Serum Magnesium; Serum Vitamin D; Serum Uric Acid
MeSH Terms: conditions — Stroke | interventions — Uric Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Serum magnesium, uric acid, and vitamin D levels and motor recovery and ambulation stages — Serum magnesium, uric acid, and vitamin D levels, as well as motor recovery and ambulation levels, measured during the patients' rehabilitation stay will be obtained from past medical records.

SUMMARY:
This study aim to retrospectively investigate the effects of the magnesium, vitamin D, and uric acid serum markers on motor recovery and ambulation in post-stroke patients.

DETAILED DESCRIPTION:
Stroke is the sudden loss of neurological function associated with a reduction or cessation of blood flow in the brain, resulting from the blockage or rupture of cerebral vessels. Stroke is the second leading cause of death and the third leading cause of disability worldwide. Regaining motor recovery and ambulation skills in patients is one of the main goals of rehabilitation. It is critical for patients to improve their quality of life and regain their independence. Serum biochemical markers can be used to predict post-stroke recovery. Serum magnesium, vitamin D, and uric acid are biochemical markers that may play a role in the recovery process of stroke patients.

This study aim to retrospectively investigate the effects of the magnesium, vitamin D, and uric acid serum markers on motor recovery and ambulation in post-stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a single stroke between 2019 and 2024
* Patients who were admitted to the rehabilitation ward and had their serum vitamin D, magnesium, and uric acid levels measured
* Patients whose functional ambulation scale scores and Brunnstrom motor recovery stages were recorded

Exclusion Criteria:

* Patients with other neurological diseases
* Patients with multiple strokes
* Patients with gout, renal failure, or hyperparathyroidism

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a stroke for the first time and are hospitalized in the rehabilitation ward for rehabilitation purposes.
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Serum magnesium levels | Before treatment
  Serum magnesium levels measured before the patients' rehabilitation will be obtained from past medical records.
Serum uric acid levels | Before treatment
  Serum uric acid levels measured before the patients' rehabilitation will be obtained from past medical records.
Serum vitamin D levels | Before treatment
  Serum vitamin D levels measured before the patients' rehabilitation will be obtained from past medical records.
Brunnstrom Motor Recovery Stage | Before treatment
  Brunnstrom stages is a scale used to assess motor recovery after a stroke, which is expressed using values between 1 and 6. The higher the value on this scale, the higher would be the recovery. Brunnstrom Motor Recovery Stages measured before the patients' rehabilitation will be obtained from past medical records.
Functional Ambulation Classification | Before treatment
  Functional Ambulation Classification is a 6-point functional walking test that evaluates ambulation ability and determines the amount of human support required by patients while walking, regardless of whether they use a personal assistive device. A score of 0 indicates that the patient has a dysfunctional ambulation A score of 5 denotes independent ambulation on any surface. Functional Ambulation Classification Stages measured before the patients' rehabilitation will be obtained from past medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided